CLINICAL TRIAL: NCT04963374
Title: Comparative Analysis of the Effectiveness of Different Risk Scales in Predicting Combined Venous Thrombophilia in Respiratory Inpatients
Brief Title: the Effectiveness of Different Risk Scales In Predicting VTE in Respiratory Inpatients
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Peking UTH
Record Dates: First submitted 2021-06-29; First posted 2021-07-15 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Venous Thromboembolism
Keywords: VTE
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- respiratory inpatient: respiratory inpatient with VTE
  Interventions: Other: risk evolution scale

INTERVENTIONS:
Other: risk evolution scale — Padua score、Caprini score、Prime score

SUMMARY:
To compare the predictive effectiveness of the Caprini risk assessment model, the Padua risk assessment model and the VTE risk assessment in medical patients mentioned in the 2018 edition of the Guidelines for the diagnosis, treatment and prevention of pulmonary thromboembolism on the risk of concomitant VTE in respiratory inpatients to provide a basis for clinical VTE assessment and treatment.

DETAILED DESCRIPTION:
A case-control study was used to collect patients who developed VTE during hospitalization in the Department of Respiratory Medicine at Peking University Third Hospital Hospital from January 2015 to December 2020 as the case group, and 2-fold patients who did not develop VTE matched to the case group (age, sex, ADL score, diagnosis, and length of hospitalization) as the control group. The general status of the patients was also assessed using the Padua risk model, the Caprini risk model, and the VTE risk assessment scale for medical patients mentioned in the 2018 edition of the Guidelines for the diagnosis, treatment, and prevention of pulmonary thromboembolism, and the relevant items involved in the assessment form were obtained by reviewing the cases.

ELIGIBILITY:
Inclusion Criteria:

* age more than 18y respiratory inpatient

Exclusion Criteria:

* Patients with deep vein thrombosis or pulmonary thromboembolism, sequelae of deep vein thrombosis, and thrombosis in other parts of lower limbs were diagnosed; Patients with severe coagulation dysfunction or other hematological diseases

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 2015 to December 2020, inpatients in respiratory department, Third Hospital of Peking University
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
VTE incidence | during hospitalization， an average of 2 weeks
  VTE incidence in patients with high risk of VTE

CONTACTS AND LOCATIONS:
Overall Officials: Jing Zhang, MD, Principal Investigator — Peking UTH
Locations (1):
- Peking UTH, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luo XY, Zhang FX. [Validation of the Caprini risk assessment model for venous thromboembolism in Chinese hospitalized patients in a general hospital]. Zhonghua Yi Xue Za Zhi. 2017 Jun 27;97(24):1875-1877. doi: 10.3760/cma.j.issn.0376-2491.2017.24.007. Chinese. PMID 28648012